CLINICAL TRIAL: NCT06019416
Title: Discrimination and Mental Health of Older Korean Adults in the U.S.: Feasibility and Pilot Trial of a Culturally Tailored Mindfulness-Positive Psychological Intervention Using Virtual Reality
Brief Title: Culturally Tailored Mindfulness-Positive Psychological Intervention Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23430
Record Dates: First submitted 2023-08-15; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Mental Health Issue
Keywords: Virtual reality; Mindfulness; Well-being; Anti-Asian Racism; Positive psychological intervention

STUDY DESIGN:
Intervention Model Description: Intervention group will receive the virtual reality-based culturally tailored mindfulness and positive psychological intervention, whereas the control group will not receive any intervention as a waitlist group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): As the intervention group, the participants should participate in three weekly scheduled mindfulness-positive psychological intervention sessions using virtual reality for 15 - 20 minutes per session.
  Interventions: Behavioral: culturally tailored mindfulness-positive psychological intervention
- Waitlist group (No Intervention): As the waitlist group, no treatment was given to the participants, while the intervention group participated in the mindfulness-positive psychological intervention for three weeks. After the three-week waiting period, the participants were contacted and asked to complete the post-measurements. After completion, the participants started with the three-week mindfulness-positive psychological intervention using virtual reality for 15 - 20 minutes. No further data was obtained from these participants after the completion of the program.

INTERVENTIONS:
Behavioral: culturally tailored mindfulness-positive psychological intervention — This 3-week culturally tailored mindfulness-positive psychological intervention instructs techniques to enhance positive emotions and meditation exercise lasting approximately 30 minutes. The culturally tailored mindfulness-positive psychological intervention consists of four modules: 1) noticing positive events, 2) amplifying positive events, 3) gratitude, and 4) mindfulness and meditation. This 3-dimensional software includes gamification features, including a virtual living room, Japanese garden, art gallery, and meditation garden.
  A private office and/or space was utilized to implement the culturally tailored mindfulness-positive psychological intervention for older Korean Americans/immigrants, provided by the recruitment sites such as non-profit organization and church. The private room at the sites had a desktop (or laptop) computer, a virtual reality device (Oculus Quest 2), a chair, and a desk.
  Arms: Intervention group

SUMMARY:
This study is to explore the experience of older Korean adults with anti-Asian racism in the U.S. and investigate the feasibility, acceptability, and preliminary efficacy of a virtual reality-based culturally tailored mindfulness-positive psychological intervention. Primary outcome is racism-related stress and secondary outcomes are negative mental health (e.g., anxiety, depressive symptoms, and anxiety) and positive psychological well-being (e.g., positive affect, optimism, life engagement, mindful attention awareness).

ELIGIBILITY:
Inclusion Criteria:

* U.S. Korean Americans/immigrants
* ≥ 60 years of age
* Korean fluency
* no medical history of cognitive impairments (e.g., dementia or Alzheimer-related diseases)
* self-reported direct experience of discrimination as per the Everyday Discrimination Scale

Exclusion Criteria:

* severe cognitive impairment denoting dementia
* other ethnicities rather than Korean Americans/immigrants
* younger than 60 years of age
* cannot speak and read Korean
* have not experienced any discrimination
* serious sensory problems negating the use of virtual reality
* medical history of epilepsy, seizures, or vertigo
* experience in mindfulness or meditation-based programs

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Racism-related stress | Pretest (baseline) and posttest (3 weeks later)
  The primary outcome is the racism-related stress measured by vicarious racism. Vicarious racism involves seven items that measure the frequency of hearing about or seeing other people of the same racial group experiencing racism: 1) in public or 2) in the news, 3) from romantic partners or, 4) friends and family members, 5) heard by politicians and 6) other public figures, and 7) seeing racist posts on social media during the Coronavirus Disease 2019 pandemic: 0 (never) - 5 (every day). Regarding racism-related stress, participants answer three questions: 1) the degree to which participants thought about these experiences (0 [never] - 4 [always]) and 2) how distressed, and 3) concerned they were about these experiences (0 [not at all] - 4 [extremely]; Cronbach's alpha = 0.89).

SECONDARY OUTCOMES:
Perceived stress | Pretest (baseline) and posttest (3 weeks later)
  Perceived stress is measured by the Perceived Stress Scale 4, which asks a 4-items about how often the participants felt or thought a certain way during the last month, given a five-point scale: 0 (never) - 4 (very often). Previous studies have indicated that internal consistency reliability of the Korean version was 0.82 (Cronbach's alpha).
Optimism | Pretest (baseline) and posttest (3 weeks later)
  Optimism is assessed using the Life Orientation Test-Revised, where respondents report their own feelings to measure individual differences in generalized optimism and pessimism. The Life Orientation Test-Revised consists of 3 optimism items, 3 pessimism items (reverse code), and 3 filler items (exclusion from the total scores. Given each item is presented on a 5-point scale (0 = I disagree a lot; 4 = I agree a lot), the total score ranges from 0 (least optimistic) to 24 (most optimistic; Cronbach's alpha = 0.72 - 0.78). Internal consistency reliability of the Korean version of the Life Orientation Test-Revised was 0.81 (Cronbach's alpha).
Positive affect | Pretest (baseline) and posttest (3 weeks later)
  Positive affect will be derived using the four positively worded items of the Center for Epidemiological Studies Depression Scale as follows: 1) I felt that I was just as good as other people, 2) I felt hopeful about the future, 3) I was happy, and 4) I enjoyed life. The sum of the four items ranges from 0 to 12. Reliability measured by internal consistency for the Korean version of the Center for Epidemiological Studies Depression Scale was 0.89 (Cronbach's alpha) in a previous publication.
Life engagement | Pretest (baseline) and posttest (3 weeks later)
  The Life Engagement Test is a 5-point Likert scale measuring participants' life engagement. The Life Engagement Test consists of six items as a continuous variable, but three items are reverse-coded so that higher scores indicate better life engagement. Possible responses for all questions are from 1 (strongly disagree) to 5 (strongly agree). There is no previous study that tested the reliability of older Korean adults. However, another study indicates a Cronbach's alpha of 0.84.
Mindful attention awareness | Pretest (baseline) and posttest (3 weeks later)
  The Mindful Attention Awareness Scale consists of 15 questions to measure dispositional mindfulness characteristics. The sample questions are: The Mindful Attention Awareness Scale is a continuous variable with response options ranging from 1 (almost always) to 6 (almost never). Previous studies used the Mindful Attention Awareness Scale for Koreans, and its internal consistency reliability ranges from 0.87 to 0.95 (Cronbach's alpha).
Everyday discrimination | Pretest (baseline)
  The Everyday Discrimination Scale measures the magnitude of unfair treatment in ongoing and routine experiences in daily life. The Everyday Discrimination Scale involves a nine-item scale with a six-point Likert scale: 0 (never) - 5 (almost every day). Its internal consistency reliability (Cronbach's alpha) according to previous studies targeting various ethnicities (e.g., White, Black, Hispanic/Latino, and Asian) was 0.88 (Cronbach's alpha).
Virtual reality safety | After every sessions (1 week later, 2 weeks later, 3 weeks later)
  The Simulator Sickness Questionnaire was developed to measure cybersickness symptoms in virtual reality research. The Simulator Sickness Questionnaire measures three domains (e.g., nausea, oculomotor, and disorientation) assessed through weighting 16 symptoms of cyber sickness. The measure is scored using a 4-point scale and weighted according to each factor to calculate the total score. Internal consistency reliability of the Simulator Sickness Questionnaire (Cronbach's alpha) was 0.94.
Technology acceptance | After every sessions (1 week later, 2 weeks later, 3 weeks later)
  Participants answer the scales involving perceived ease of use, perceived usefulness, and attitude toward using virtual reality, with a 5-point Likert scale (1: strongly disagree; 5: strongly agree).
Patient-Reported Outcomes Measurement Information System Bank v1.0 - Anxiety | Pretest (baseline) and posttest (3 weeks later)
  The Patient-Reported Outcomes Measurement Information System Bank v1.0 - Anxiety consists of 4 questions to measure anxiety levels. This measurement ranges from 1 (never) to 5 (always).
Patient-Reported Outcomes Measurement Information System Bank v1.0 - Depression | Pretest (baseline) and posttest (3 weeks later)
  The Patient-Reported Outcomes Measurement Information System Bank v1.0 - Depression consists of 4 questions to measure depressive symptom levels. This measurement ranges from 1 (never) to 5 (always).

OTHER OUTCOMES:
Demographic variables | Pretest (baseline)
  Demographic variables include age, sex, income level, years living in the U.S., education years, employment status, marital status, and health insurance.
Intervention feasibility | posttest (3 weeks later)
  Feasibility consists of recruitment rates (potential participants who were approached for recruitment), enrollment rates (≥20% of participants who decide to enroll), retention/attrition rates (goal: 70% of participants who completed the post-intervention assessment, answering Yes/No), and (non)compliance or adherence rates.

CONTACTS AND LOCATIONS:
Overall Officials: Soonhyung Kwon, MSW, MA, Principal Investigator — University of Illinois Urbana-Champaign, School of Social Work
Locations (3):
- United States (3):
  - Xilin Association, Chicago, Illinois
  - Hanul Family Alliance, Chicago, Illinois
  - Christ Community Church at the Square, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No
This is a dissertation project. This study data will not be shared with other researchers